CLINICAL TRIAL: NCT07270640
Title: Lifestyle Intervention to Improve Twin Pregnancy Outcomes: an Integrated Pilot Study for a Multicentric Randomized Controlled Trial
Brief Title: Lifestyle Intervention to Improve Twin Pregnancy Outcomes
Acronym: LIFETWIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S68251
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Twin Pregnancy, Dichorionic
Keywords: twin pregnancy; dichorionic; lifestyle interventions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Lifestyle coaching sessions
  Interventions: Behavioral: LIFETWIN
- Control (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: LIFETWIN — The LIFETWIN intervention provides 8 coaching sessions to women during pregnancy, focusing on nutrition (including multivitamin intake), physical activity and stress reduction.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial to is assess the benefits of holistic lifestyle interventions, including nutrition, physical activities, and mindfulness, aiming to reduce preterm birth in twins, potentially revolutionizing twin care globally.

An initial integrated pilot study is be conducted to assess and refine the intervention methods. The primary objective of the pilot study is to evaluate feasibility. If deemed feasible, the full study will be implemented, incorporating data from pilot study participants into the main study.

Objective of the full study: To evaluate if a multi-component lifestyle extends gestational age at delivery by one week. Additional objective: to evaluate if the intervention positively influences multiple secondary outcomes including pregnancy complications, neonatal and maternal outcomes, and maternal quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Prior to any randomization or intervention, participants must have provided voluntary written informed consent.
* Diagnosis of dichorionic twin pregnancies must align with the acceptance criteria.
* Participants must be recruited before the 14th week of gestation.
* Proficiency in Dutch, English, or French is required.-

Exclusion Criteria:

* Participant has a history of pre-existing diseases or condition impacting their diet:

  1. pre-gestational diabetes
  2. severe heart disease,
  3. chronic renal disease,
  4. celiac disease,
  5. inflammatory bowel disease,
  6. post-bariatric surgery
* Participant has a history of pre-existing diseases or conditions impacting their physical activity ability:

  1. Chronic Obstructive Pulmonary Disease (COPD)
  2. Severe Asthma.
  3. Fibromyalgia
  4. Osteoarthritis
  5. Chronic Pain Syndromes
  6. Spinal Cord Injuries.
  7. Multiple Sclerosis (MS)
  8. Parkinson's Disease
  9. History of a Stroke
  10. Drug resistance Epilepsy
* Participants identified with mental vulnerabilities requiring specific care pathways by Born in Belgium (BIB) or local screening tool.
* Participants with a History of Mental Health Disorders

  1. Post-Traumatic Stress Disorder (PTSD)
  2. Anxiety Disorders
  3. Depressive Disorders
  4. Bipolar Disorder
  5. Obsessive-Compulsive Disorder (OCD)
  6. Schizophrenia or schizoaffective disorder
* Inability to give informed consent
* No knowledge of Dutch, English or French
* First trimester diagnosis of severe congenital anomaly in one or both twins
* First trimester foetal demise of one or both twins
* Rupture of membranes prior to recruitment
* Participation in any other interventional Study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Gestational age at delivery | Delivery
  The primary outcome is gestational age at delivery, measured in weeks and days. This is calculated based on the last menstrual period and confirmed via early ultrasound dating (before 13 weeks and 6 days) for spontaneous pregnancies or based on embryo age at transfer for IVF patients. The study aims to evaluate whether a multi-component lifestyle intervention can delay delivery by at least one week, thereby enhancing pregnancy outcomes. Gestational age data will be collected from medical records to ensure accuracy and consistency.

SECONDARY OUTCOMES:
Birth weight | Delivery
  Birth weight in grams and percentile.
Small for gestational age | Delivery
  Small for gestational age in at least one twin, defined as below the 10th percentile according to twins' nomograms
Offspring mortality | 24 weeks -28 days postpartum
  Offspring mortality- defined as the death of one or both twins occurring at any time from foetal viability (24 weeks' gestation) until 28 days postpartum (neonatal period).
Offspring infection | within the first 72 hours of delivery
  Offspring infection- defined as neonatal sepsis, congenital pneumonia, neonatal meningitis, or necrotizing enterocolitis (NEC) with infection within the first 72 hours of delivery.
Early neurodevelopmental morbidity | 6 weeks postpartum
  Early neurodevelopmental morbidity- defined as diagnosis of Intraventricular haemorrhage (IVH) Grade III-IV, periventricular leukomalacia (PVL), hypoxic-ischemic encephalopathy (HIE), and neonatal seizures.
Gastrointestinal morbidity | 6 weeks postpartum
  Gastrointestinal morbidity- defined as diagnosis of NEC and spontaneous perforation.
Respiratory morbidity | 6 weeks postpartum
  Respiratory morbidity- defined as diagnosis of respiratory distress syndrome (RDS), bronchopulmonary dysplasia (BPD), transient tachypnoea of the newborn (TTN) or persistent pulmonary hypertension of the newborn (PPHN)
NICU admission | within 72 hours of delivery
  Any admission to the Neonatal intensive care unit (NICU) within 72 hours of delivery.
Number of days in the NICU | 6 weeks postpartum
  Number of days in the NICU
Gestational weight gain | from 14 weeks pregnancy to delivery
  Gestational Weight Gain (GWG) corrected to pregnancy duration.
Maternal quality of life | Before 14 weeks of pregnancy, 32-34 weeks and 6 weeks postpartum
  Maternal quality of Life based on questionnaire EQ-5D-5L.
Postpartum weignt | 6 weeks postpartum
  Postpartum weight recorded 6 weeks postpartum

OTHER OUTCOMES:
Maternal mortality | within 42 days postpartum
  Maternal mortality- defined as death of the mother during pregnancy or within 42 days postpartum, due to any cause related to or aggravated by pregnancy or its management.
Caesarean section delivery | delivery
Premature rupture of the membranes | before week 34
Maternal number of days in hospitalization after delivery. | 6 weeks postpartum
Maternal pregnancy related hypertension | from 14 weeks of pregnancy to delivery
  Maternal pregnancy related hypertension- defines as Pregnancy-induced hypertension or preeclampsia as defined by the International Society for the Study of Hypertension in Pregnancy (ISSHP).
Maternal gestational diabetes mellitus | from week 20 of pregnancy to delivery
  Maternal gestational diabetes mellitus as defined by diagnosis of diabetes after week 20 in a two-step approach according to the Carpenter/Coustan criteria.
maternal anaemina | from 14 weeks of pregnancy to delivery
  Maternal anaemia defined by haemoglobin under 10 g/dL during pregnancy.
Food consumption change | before 14 weeks, 32-34 weeks of pregnancy and 6 weeks postpartum
  Food consumption change based on 32-item semi-quantitative Food Frequency Questionnaire
Physical activity | before 14 weeks, 32-34 weeks, 6 weeks postpartum
  Physical activity level based on the Kaiser Physical Activity Survey.
Change in lifestyle habits | before 14 weeks, 32-34 weeks, 6 weeks postpartum
  Change in lifestyle habits based on Lifestyle behaviour questionnaire.
Neonatal number of days in hospitalization after delivery. | 6 weeks after birth
Number of recruited participants | through study completion, an average of 1.5 years
  Recruitment Success (RE-AIM Principle: Reach and Adoption): assessment the ability to recruit participants over the course of the pilot. Recruitment efforts will focus on engaging a diverse demographic, particularly including women from low SES and high-risk backgrounds.
Training and retention of study midwifes | through study completion, an average of 1.5 years
  Midwife Engagement (RE-AIM Principle: Adoption): Midwives at all centres will undergo a two-day training program tailored to the LIFETWIN intervention. Retention and engagement of midwives will be monitored throughout the study.
Consistency of intervention delivery | through study completion, an average of 1.5 years
  Intervention Fidelity (RE-AIM Principle: Implementation): We will assess how consistently the intervention (8 lifestyle sessions) can be delivered, both face-to-face and remotely, ensuring quality and adherence across both centres.
The number of participants retained throughout the pilot study | through study completion, an average of 1.5 years
  Participant Retention (RE-AIM Principle: Maintenance): Monitor retention rates of participants throughout the study period, with reasons for lack of adherence and dropout carefully recorded. This will help us understand both the feasibility of maintaining participant engagement and the practical challenges in long-term implementation
Qualitative feedback on experiences with the intervention | through study completion, an average of 1.5 years
  Qualitative Feedback (RE-AIM Principle: Maintenance): Midwives and participants will be interviewed to assess how the intervention is perceived, experienced, and sustained over time. Insights from this feedback will be critical for informing the next phase of the study, especially regarding long-term adoption and sustainability.

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - CHU Brugmann, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Leuven, Leuven
  - Hôpital de la Citadelle, Liège

IPD SHARING:
Plan to Share IPD: Undecided